CLINICAL TRIAL: NCT06118788
Title: A Single-arm, Dose-escalation and Dose-expansion Phase I Clinical Study to Evaluate the Tolerability, Safety and Preliminary Efficacy of BG1805 Injection in the Treatment of Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Phase I Clinical Study: BG1805 Injection in the Treatment of Relapsed or Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangzhou Bio-gene Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG-CA-22-001
Record Dates: First submitted 2023-10-30; First posted 2023-11-07 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: CAR-T; AML; CLL1
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BG1805 (Experimental): Dose escalation: Three dose levels were designed, and if the maximum tolerated dose (MTD) was not found at the highest level, no further dose escalation was to be performed. Approximately 12-18 subjects were planned to be enrolled in the dose-escalation phase to evaluate the safety and tolerability of BG1805 injection and to determine the MTD and/or the recommended phase II dose (RP2D).
  Dose Expansion: During or after the dose escalation process, if a certain dose group is determined to have preliminary anti-tumor effects and controllable safety, it can be extended at this dose level to further evaluate the tolerance and safety of BG1805 injection, and to preliminarily evaluate its effectiveness.
  Interventions: Biological: BG1805

INTERVENTIONS:
Biological: BG1805 — A single infusion of BG1805 Injection administered intravenously.

SUMMARY:
This is a single-arm, single-dose dose-escalation and dose-expansion study.

DETAILED DESCRIPTION:
Patients with relapsed/refractory acute myeloid leukemia (r/r AML) were enrolled in the trial, which was divided into two parts: dose-escalation phase and dose-expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent and be expected to complete the follow-up examination and treatment of the study procedures.
2. Age of 18-70 years old (inclusive of the cut-off value), regardless of gender.
3. Conforming to the diagnosis of AML according to the 2016 WHO classification, and conforming to the diagnostic criteria of relapsed and refractory acute myeloid leukemia in Chinese Guidelines for the Diagnosis and Treatment of relapsed and refractory acute myeloid Leukemia (2017 edition) :

   1. Relapsed AML diagnostic criteria: the reappearance of peripheral blood or bone marrow blasts after complete remission (CR); 5% (excluding other causes such as bone marrow regrowth after consolidation chemotherapy) or extramedullary leukemic cell infiltration.
   2. Refractory AML diagnostic criteria: newly diagnosed patients who failed to response to 2 courses of standard regimens; Patients who relapsed within 12 months after consolidation and intensive therapy; Patients relapsed after 12 months but failed to respond to conventional chemotherapy; Patients with two or more recurrences; Patients with persistent extramedullary leukemia.
4. Flow cytometry confirmed the AML Blast CLL-1 expression positive (CLL-1 expression ≥50%).
5. The patient has recovered from the toxicity of previous treatment, defined as CTCAE toxicity grade <2 (unless the abnormality is tumor-related or is judged by the investigator to be stable and has little effect on safety or efficacy).
6. ECOG performance status of 0-1 and predicted survival of more than 3 months.
7. Have appropriate organ functions:

   * Aspartate aminotransferase (AST) ≤3 times the upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) ≤3 times ULN
   * Total bilirubin ≤1.5 times ULN
   * Serum creatinine ≤1.5 times ULN or creatinine clearance ≥60 mL/ minute
   * Hemoglobin ≥60g/L or maintained at that level after transfusion
   * Refers to terminal oxygen saturation ≥92%
   * Left ventricular ejection fraction (LVEF) ≥45%
8. Female subjects were also considered for inclusion if they met the following criteria:

   1. Infertility, defined as:

      * Prior hysterectomy or bilateral oophorectomy, or
      * Prior bilateral tubal ligation, or
      * Menopausal (≥ 1 year of complete amenorrhea)
   2. be fertile, but have a negative serum pregnancy test at screening, and agree to use a medically approved contraceptive method (e.g., an intrauterine device, contraceptive pill, or condom) before and during study enrollment and up to 1 year after the last study use.
9. Men of childbearing potential had to agree to barrier contraception or complete abstinence until 1 year after the last study dose.

Exclusion Criteria:

1. Acute promyelocytic leukemia was diagnosed.
2. Have other malignant tumors within 3 years before screening, excluding adequately treated cervical carcinoma in situ, papillary thyroid carcinoma, basal cell or squamous cell skin cancer, local prostate cancer after radical prostatectomy, and ductal carcinoma in situ after radical prostatectomy.
3. Evidence of central nervous system involvement or cranial neuropathy.
4. Hepatitis B surface antigen (HBsAg) positive, hepatitis B core antibody (HBcAb) positive and peripheral blood HBV-DNA higher than the detection limit; Hepatitis C virus (HCV) antibody positive; Persons with human immunodeficiency virus (HIV) antibody positive; Cytomegalovirus (CMV) DNA positive cases; EBV-DNA positive patients; The syphilis antibody was positive.
5. Those with a history of anaphylaxis [A history of anaphylaxis was defined as an allergic reaction of grade 2 or higher, in which any of the following clinical manifestations occurred: Airway obstruction (rhinorrhea, cough, stridor, dyspnea), Tachycardia, Hypotension, Arrhythmia, Gastrointestinal symptoms (nausea, vomiting), Incontinence, Laryngeal edema, Bronchospasm, Cyanosis, Shock, Respiratory, cardiac arrest] or known to be allergic to any of the drug active ingredients, excipents, or mouse-derived products or xenoproteins included in this trial (including the lymphatic cells clearance protocol).
6. Have severe cardiac disease, including but not limited to severe arrhythmia, unstable angina, massive myocardial infarction, New York Heart Association class III or IV cardiac dysfunction, and refractory hypertension.
7. Previous organ transplantation or preparation for organ transplantation (excluding hematopoietic stem cell transplantation).
8. Acute and chronic graft-versus-host disease (GVHD).
9. Patients who had undergone hematopoietic stem-cell transplantation within 6 months before screening.
10. Active autoimmune or inflammatory diseases (e.g., Guillain-Barre syndrome (GBS), amyotrophic lateral sclerosis (ALS)) and clinically significant active cerebrovascular diseases (e.g., cerebral edema, posterior reversible encephalopathy syndrome (PRES)).
11. Patients with cancer emergencies (such as spinal cord compression, intestinal obstruction, leukostasis, tumor lysis syndrome, etc.) requiring emergency treatment before screening or reinfusion.
12. Presence of uncontrolled bacterial, fungal, viral, or other infection requiring antibiotic treatment.
13. Patients who had undergone major surgery (excluding diagnostic surgery and biopsy) within 4 weeks before lymphatic cells clearance or planned to undergo major surgery during the study period, or who had not fully healed the surgical wound before enrollment.
14. Persons with severe mental illness.
15. Within 1 week before the collection of peripheral blood mononuclear cells (PBMC), patients who use granulocyte colony-stimulating factor (G-CSF), granulocyte macrophage colony-stimulating factor (GM-CSF) and other hematopoietic cytokine drugs that have an impact on the patient's blood picture (if it is a long-acting preparation, it is 2 weeks) and have an impact on cell preparation as judged by the investigator .
16. Within 2 weeks before PBMC collection, patients were receiving hormonal or immunosuppressive drugs that were judged by the investigator to have an effect on cell production.

    1. hormone: subjects who were receiving systemic steroid therapy within 2 weeks before PBMC collection and who required long-term systemic steroid therapy (except inhaled or topical use) as judged by the investigator during the treatment.
    2. Immunosuppressive agents: those who were receiving immunosuppressive agents within 2 weeks before PBMC collection.
17. Vaccination with live (attenuated) virus vaccine within 4 weeks prior to screening.
18. Alcoholics or those with a history of substance abuse.
19. Participate in other clinical investigators within 3 months.
20. Subjects who have received other CAR-T therapy or cell therapy in the past.
21. Patients who, in the investigator's judgment and/or clinical criteria, have contraindications to any study procedure or other medical conditions that may put them at unacceptable risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity Rate | Up to 28 days after BG1805 infusion.
  After the infusion of BG1805, subjects still experienced adverse events, meeting the DLT definition, related to or possibly related to BG1805 infusion after optimal supportive treatment.
Incidence of Treatment-Emergent Adverse Events | Up to 24 months.
  Count the Incidence of adverse events.

SECONDARY OUTCOMES:
Concentration of CAR-T cells after Infusion (PK) | Up to 24 months.
  CAR-T in peripheral blood after infusion
overall response rate, ORR | Up to 24 months.
  Defined as the proportion of subjects achieving complete response(CR), complete remission with incomplete blood cell recovery (CRi), morphologic leukemia-free state (MLFS), or partial response(PR).
Concentration of Cytokine after Infusion (PD) | Up to 24 months.
  Calculate the change of cytokine concentration in peripheral blood after After BG1805 infusion. Cytokines include IL-2、IL-6 and so on.

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — Zhejiang University
Locations (3):
- China (3):
  - ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang